CLINICAL TRIAL: NCT01865643
Title: A Comparison of Two GlideScope Intubation Techniques - Effect on Hemodynamic Changes and Injury Rate
Brief Title: A Comparison of Two GlideScope Intubation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-03
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Intubation, Endotracheal; Anesthesia, General
Keywords: Laryngoscopy; Intubation; Glidescope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard GlideScope intubation (Other): This standard GlideScope (GS) technique involves a midline larygoscopy followed by insertion of a styleted endotracheal tube, once an adequate view of the vocal cords is achieved.
  Interventions: Device: GlideScope
- Alternative GlideScope intubation (Experimental): Alternative GlideScope (GS) intubation involves the insertion of the endotracheal tube under direct vision as a "fish hook" at the side of the mouth before the GS blade is introduced into the oropharynx.
  Interventions: Device: GlideScope

INTERVENTIONS:
Device: GlideScope — The GlideScope is used to assist with difficult tracheal intubation.

SUMMARY:
The aim of this study is to compare the hemodynamic response to tracheal intubations using the standard technique versus the alternative GS intubation technique. As secondary outcomes the investigators will analyze procedure time, success rate and injury rate.

The investigators hypothesize that the alternative intubation technique will have a shorter procedure time and lower injury rate when compared to the standard technique of GS intubation.

DETAILED DESCRIPTION:
A Difficult intubation is still one of the most daunting challenges in anesthesiology. One of the tools used to assist with a difficult tracheal intubation is the GlideScope (GS) (Verathon, Bothell, WA, USA). The GS is a video laryngoscope that has a 60 degree angle blade with a built-in high-resolution camera and a light source assembled beside it. The image is transmitted onto a mobile bedside monitor. It has been widely used in medicine for over a decade. The GS was designed to provide an improved view of the glottis during difficult intubations without alignment of the oral, pharyngeal and tracheal axes, as it is able to "look around the corner" to facilitate the intubation.

The standard technique of the GS intubation involves a midline laryngoscopy followed by the insertion of a styleted endotracheal tube (ETT) once an adequate view of the vocal cords has been achieved. The ETT insertion process requires the operator to look away from the monitor during the laryngoscopy while maintaining the blade position in order to insert it into its initial position.

An alternative GS intubation technique has been described for cases in which there is limited mouth opening, a big tongue or other anatomical impediments. In these cases the ETT is inserted under direct vision as a "fish hook" at the side of the mouth before the GS blade is introduced into the oropharynx.

There are several advantages to this alternative technique. The first advantage is that this technique of ETT insertion would minimize the laryngoscopy time as a part of it is performed before the blade is introduced and the stimulating effect occurs. This technique thus has the potential of reducing the sympathetic response. Minimizing oropharyngo-laryngeal stimulation time would theoretically attenuate the hemodynamic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA physical status 1-2
* Patients aged 18 years and older
* Patients undergoing elective surgery that requires tracheal intubation

Exclusion Criteria:

* Patients in whom a rapid sequence intubation or alternative intubation method is indicated
* Patients with a known or suspected oral, pharyngeal or laryngeal mass
* Patients previously flagged as a difficult intubation
* Patients with hypertension (treated or untreated, poor dentition, symptomatic gastro-esophageal reflux or cervical spine instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hemodynamic response to tracheal intubation | 24 hours
  Heart rate and non-invasive blood pressure will be measured before induction, and throughout and after laryngoscopy and induction

SECONDARY OUTCOMES:
Procedure time | 10 minutes
  Time for intubation will be measured as time from laryngoscopy to the inflation of the ETT cuff.
Success rate | 10 minutes
  Successful placement of endotracheal tube between the vocal cords.
Injury rate | 30 minutes
  Injuries to the oropharynx

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Friedman, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada